CLINICAL TRIAL: NCT02256020
Title: Improvement and Mechanism of Wheel-chair Music Aerobic Exercise on Depression and Insomnia Among the Elderly in Long-term Care Facilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-Hui Yeh, RN, PhD, Professor, Chang Bing Show Chwan Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1030104
Record Dates: First submitted 2014-09-24; First posted 2014-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Wheel-chair Dependent Elders
Keywords: Wheel-chair dependent, music aerobic exercise, depression, insomnia
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Original lifestyle (Other): Original lifestyle, watching TV 50 minutes, three times a week for 6 months.
  Interventions: Other: Original lifestyle
- Wheel-chair music aerobic exercise (Experimental): Wheel-chair music aerobic exercise with 3 times of 50-minute session (10 minutes warm up, 30 minutes exercise and 10 minutes cool down) a week for 6 months.
  Interventions: Other: Wheel-chair music aerobic exercise (WC-MAE)

INTERVENTIONS:
Other: Original lifestyle — Control group with 3 times of watching 50-minute television a week for 6 months.
  Arms: Original lifestyle
Other: Wheel-chair music aerobic exercise (WC-MAE) — Wheel-chair music aerobic exercise with 3 times of 50-minute session a week for 6 months.
  Arms: Wheel-chair music aerobic exercise

SUMMARY:
Investigators anticipate to develop a customized WC-MAE for the improvement of insomnia and depression in wheel-chair dependent elders, and to identify related mechanisms as biomarkers for prediction and prevention of insomnia and depression in elders with physical disability in long term care facilities.

DETAILED DESCRIPTION:
It has been shown that two-thirds of elderly residents living in long term care facilities lack regular exercise. The lack of physical activity may cause decreased physical function, impaired immunity, insomnia and depression. Insomnia can affect circadian rhythm, control of emotion and blood pressure. Depression can affect hormone regulation and quality of life. More importantly, depression has been recognized as one of the world's top three health problems by the World Health Organization. In Taiwan, our previous study showed that the prevalence of depression in community elderly was 27.5% (Tsai, Yeh & Tsai, Int J Geriatric Psychiatr. 2005). We also demonstrated that Tai Chi Chuan exercise improved balance, nerve conductivity and immunity (Yeh, Chuang, Lin, Hsiao, & Eng, Br J Sports Med. 2006; Hung, Liou, Wang, & Yeh, J Rehabilit Med. 2009). A recent study that followed 3500 elders (> 64 years of age) for 8 years in the United Kingdom showed that exercise, no matter at what age it began, significantly improved physical function (Kaasalainen, Kasila, Villberg, Komulainen, & Poskiparta, BMC Public Health. 2013). Thus, we hypothesized that those wheel-chair dependent elders, who exercise less due to physical disability, have poor sleep quality that causes emotional disturbance and potential depression. A customized wheel-chair exercise for the elderly of long term care facilities might promote physical activity and improve insomnia and depression.

Tai-chi Chuan exercise requires more endurance of static posture and is not suitable for wheel-chair dependent elders. Our preliminary studies have found that music aerobic exercise (MAE) could enhance certain immune functions of middle-age women (Yeh, Lai, Hsiao, Lin, Chung, & Yan, J Phys Act Health 2013). We chose to modify the MAE to a customized wheel-chair music aerobic exercise (WC-MAE) for physical disabled elders in long term care facilities. During the past year, we have effectively modified the original MAE to be a novel WC-MAE. We developed a WC-MAE program consisting of three weekly 50 minute sessions. These sessions are classified as moderate exercise with a goal of a maximum heart rate (HRmax) of 65%. During this 2-year project, we will do cluster randomization of 170 participants (85 pairs) from 4 long term care facilities into experimental group (with WC-MAE at 10 minutes warm up, 30 minutes exercise and 10 minutes cool down) and comparison group (watching TV 50 minutes), based on the power of 0.8, effect size of 0.28, one-tailed, alpha value of 0.05 and 10% withdrawal rate. In the first year, we will examine the effects of WC-MAE on wheel-chair dependent elders on self-perceived health, outcome expectation of exercise, and improvement of insomnia and depression scores, in pretest and the posttest at 3 months. During the second year we will study the post-test at 6 months, and investigate the mechanisms of the improvement on insomnia and depression. Blood leukocytes and plasma will be collected at pre-test, 3 and 6 months post-test for investigating changes of circadian gene expression, inflammatory cytokines, and neuro-related hormones in leukocytes and plasma. The circadian rhythm, immunity and hormone pathways will be analyzed and correlated to changes in the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Live in central and southern Taiwan
* Resident in one of the selected long-term care facilities and age 65 years or above
* Able to communicate in Mandarin or Taiwanese

Exclusion Criteria:

* Severe cognitive deficit (screen by using short portable mental status questionnaire, SPMSQ) (Pfeiffer, 1975)
* Major cardiovascular diseases, requires screening before the exercise
* Immune diseases
* Drug-induced depression

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Phenotype improvement | Change from baseline in phenotype at 6 months
  The participants will receive depression and insomnia measured before exercise and at 3 months and 6 months after starting WC-MAE to detect the changes of outcome indicators. The structured questionnaire interview will be done in each participant's long term care facilities by clinical study nurses. Five structured questionnaires including Short Portable Mental Status Questionnaire (SPMSQ) (Pfeiffer, 1975), demographic questionnaire, Beck Depression Inventory II (Bect, Steer & Brown, 1996), Pittsburgh Sleep Quality Index, (PSQI) (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989) and Outcome Expectation for Exercise (OEE) will be used for data collection.

SECONDARY OUTCOMES:
Changes of neuro-related hormones | Changes from baseline in neuro-related hormones at 6 months
  Peripheral blood will be collected before exercise and at 3 months and 6 months after starting WC-MAE to detect the changes of neuro-related hormones including DHEA-S, estradiol, DHT, progesterone, pregnenolone, total and free testosterone, epinephrine, norepinephrine, BDNF and GH.
Changes of circadian gene expression | Changes from baseline in circadian gene expression at 6 months
  Peripheral blood will be collected before exercise and at 3 months and 6 months after starting WC-MAE. After separation of blood leukocytes, the total RNA will be extracted to detect the changes of circadian gene expression including PER1, DBP, NR1D1, BMAL.
Immune function improvement | Changes from baseline in immune function at 6 months
  Peripheral blood will be collected before exercise and at 3 months and 6 months after starting WC-MAE to detect the changes of lymphocyte subpopulations (Th1/ Th2/ Treg/ Th17), polarization (T-bet/ Gata-3/ Foxp3/ RORrt), its related cytokines (Th1: IL-12/ IFN-γ/ IL-27; Th2: IL-4/ IL-13/ IL-25; Th17: IL-17A/ IL-6/ IL-21; Treg: TGF/ IL-10).

CONTACTS AND LOCATIONS:
Overall Officials: Kuender D. Yang, PhD, Study Chair — Chang Bing Show Chwan Memorial Hospital; Shu-Hui Yeh, PhD., Principal Investigator — Chang Bing Show Chwan Memorial Hospital & Central Taiwan University of Science and Technology; Li-Wei Lin, PhD, Principal Investigator — Department of Nursing, Hung Kuang University; Yu-Guan Zhuang, M.S.N, Principal Investigator — Yin Huo Health Association
Locations (1):
- Division of Core Laboratory; Chang Bing Show Chwan Memorial Hospital, Changhua County, Taiwan